CLINICAL TRIAL: NCT00798265
Title: A Phase I Study of Quadrivalent Human Papilloma Virus (HPV) (Types 6, 11, 16, 18) Recombinant Vaccine in HIV-Infected and HIV-Negative Pre-Adolescents, Adolescents and Young Adults
Brief Title: A Phase I Study of Quadrivalent Human Papilloma Virus (HPV) (Types 6, 11, 16, 18) Recombinant Vaccine in HIV-Infected and HIV-Negative Pre-Adolescents, Adolescents, and Young Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to low accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hoyoung M. Maeng, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 090024; 09-C-0024
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Human Immunodeficiency Virus; Human Papillomavirus- 6, 11, 16, 18; Adolescent; Papillomavirus Vaccines
Keywords: HPV Vaccination; HPV Immunogenicity; HIV Infection; HIV Negative; Adolescents and Young Adults; Healthy Volunteer; HV; Adolescent
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Human Papillomavirus Recombinant Vaccine nonavalent; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 - 0.5 mL dose injected intramuscular (IM) (Experimental): 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0
  Interventions: Biological: Gardasil; Behavioral: Survey
- Cohort 2 - 0.5 mL dose injected intramuscular (IM) (Experimental): 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0
  Interventions: Biological: Gardasil; Behavioral: Survey
- Cohort 3 - 0.5 mL dose injected intramuscular (IM) (Active Comparator): 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0
  Interventions: Biological: Gardasil; Behavioral: Survey

INTERVENTIONS:
Biological: Gardasil — .5 mL dose injected intramuscular (IM) at 0, 2 and 6 months
  Other Names: Human Papillomavirus 9-valent Vaccine, Recombinant
Behavioral: Survey — Administration of online risk behavior and knowledge survey done at week 0.

SUMMARY:
Background:

* Human papilloma virus (HPV) is a common sexually transmitted disease. There are more than 100 different HPV types, and both males and females can get HPV infection. Most people do not have any symptoms when they become infected and are able to get rid of the infection on their own. However, they can still become re-infected with the same or a different HPV type, and in some people HPV infection persists.
* Persistent HPV infection is associated with the development of precancerous lesions and cancer. HPV types are classified as either high risk or low risk based on whether their persistence will lead to cancer.
* Patients who have suppressed immune systems are at a higher risk for HPV-related complications. They are more likely to contract multiple HPV types and have more persistent infection that can lead to precancerous lesions or cancer, which are then difficult to treat and often recur.
* A recently approved vaccine for HPV induces immunity to HPV 6, 11, 16, and 18. It was shown to be highly effective in preventing infection with these HPV types, and is approved for use in females 9 to 26 years of age. However, much less is known about the vaccines ability to induce immunity in males or individuals with suppressed immune systems.

Objectives:

- To investigate whether the HPV vaccine is safe to give and able to induce immunity in both female and male adolescents and young adults with HIV infection compared to healthy, human immunodeficiency virus (HIV)-negative persons of the same age.

Eligibility:

- Males and females, 12 to 26 years of age, divided into three groups: (1) Healthy and HIV-negative, (2) HIV-positive and on antiretroviral therapy, and (3) HIV-positive and not on antiretroviral therapy.

Design:

* Before beginning vaccination, participants will have a complete physical examination and blood drawn for routine blood tests, special tests of the immune system, antibody tests, and an HIV test.
* HPV vaccine will be given by injection into the muscle at 0, 2, and 6 months, according to the standard vaccination schedule.
* Patients with HIV infection will be monitored for a week following the first injection to test the level of HIV in the blood 3 days and 5 days after the first injection.
* Participants will also be asked to fill out a 10- to 15-minute Web-based survey about awareness, health behaviors, and personal choices related to risk factors for HIV, HPV, and other sexually transmitted diseases. Participants are not required to fill out the survey to receive the vaccine.
* The total duration of the study is 4 years. During the first year of the study, participants will return for six additional 1-day visits at months 1, 2, 3, 6, 7, and 12. Participants will return for 1-day visits every 6 months for the remaining 3 years.

DETAILED DESCRIPTION:
Background:

Human papilloma virus (HPV) is one of the most common sexually transmitted diseases and a significant cause of cutaneous genital warts and anogenital cancer.

Infection with high-risk, oncogenic HPV types, most commonly types 16 and 18, is associated with low and high-grade cervical cellular abnormalities that are precursors to invasive cervical cancer, as well as vulvar and anal cancer, while HPV types 6 and 11 are associated with genital warts.

Persistence of HPV infection is more common in individuals with or at risk for chronic immunosuppression and HIV-infected individuals have a higher prevalence of HPV infection and HPV-associated anogenital disease compared to age-matched human immunodeficiency virus (HIV)-negative controls.

Study Objectives:

To assess the safety and immunogenicity of quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine in HIV-infected preadolescents, adolescents and young adults 12-26 years of age.

To determine whether there are differences in HPV vaccine immunogenicity between HIV-infected and HIV negative age-matched controls.

To determine whether there are differences in HPV vaccine immunogenicity between HIV-infected patients receiving highly active antiretroviral therapy (HAART) and those not receiving HAART with similar cluster of differentiation 4 (CD4) and viral load parameters at entry.

To determine whether HPV vaccination alters human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) levels.

To investigate the impact of CD4 count and HIV-1 RNA levels on HPV vaccine immunogenicity.

To characterize HPV deoxyribonucleic acid (DNA) positivity in the study cohort populations through oral/buccal and anogenital sampling at baseline.

To characterize HPV and HIV knowledge and risk and sexual behaviors in the study cohort populations.

Eligibility:

Individual Cohorts

Cohort 1: HIV-positive, CD4 cell count greater than or equal to 350 cells/mm^3, HIV-1 RNA level by reverse transcription (RT) polymerase chain reaction (PCR) less than or equal to 20,000 copies/ml, on stable HAART regimen for greater than or equal to 6 months.

Cohort 2: HIV-infected, CD4 cell count greater than or equal to 500 cells/mm^3, HIV-1 RNA level by RT PCR less than or equal to 20,000 copies/ml, on no antiretroviral treatment.

Cohort 3: healthy, HIV-negative controls All Cohorts

Females and males age 12 to 26 years

Patients must have a hemoglobin greater than or equal to 10.0 gm/dL, neutrophil count (ANC) greater than or equal to 1500/mm^3, platelet count greater than or equal to 75,000/mm^3 and prothrombin time (PT) or partial thromboplastin time (PTT) less than or equal to 1.5x upper limit of normal (ULN) (with the exception of patients with known clotting disorders or lupus anticoagulant); serum glutamic-pyruvic transaminase (SGPT)/Serum glutamic oxaloacetic transaminase (SGOT) < 2/5x ULN, total bilirubin less than or equal to 1.5x ULN unless attributable to protease inhibitor therapy.

Patients must test negative for hepatitis B virus and hepatitis C virus, unless the result is consistent with prior vaccination or prior infection with full recovery.

No use of investigational agents within 4 weeks of study enrollment or use of immunosuppressive or immunomodulating agents within 8 weeks of study entry.

Study Design:

This is a non-randomized, prospective, phase I study of quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine.

The study includes 3 cohorts of pre-adolescents, adolescents and young adults 12-26 years of age as outlined under Eligibility Criteria. Each cohort will enroll 35 patients.

All study subjects will receive three doses of HPV vaccine at 0, 2 and 6 months administered IM.

Study participants will be monitored at months 0, 1, 2, 3, 6, 7, and 12 (+/- 2 weeks for each visit, and every 6 months (+/- 30 days) thereafter for 48 months total.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Cohort 1 Inclusion and Exclusion Eligibility Criteria:

INCLUSION CRITERIA:

2.1.1.1 Age 12 to 26 years

2.1.1.2 Females and males

2.1.1.3 Human immunodeficiency virus (HIV)-positive

2.1.1.4 Cluster of differentiation 4 (CD4) cell count and Human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) level parameters

* CD4 cell count greater than or equal to 350 cells/mm(3)
* HIV-1 RNA level by reverse transcription-polymerase chain reaction (RT PCR) less than or equal to 20,000 copies/ml

2.1.1.5 On stable highly active antiretroviral therapy (HAART) regimen for greater than or equal to 6 months with CD4 and viral load parameters as outlined in 2.1.1.4

2.1.1.6 Patients greater than or equal to 18 years willing to provide informed consent or parent/guardian willing to provide informed consent for minor children less than 18 years of age.

2.1.1.7 Informed assent for patients 12-17 years of age (Optional at the discretion of the Principal Investigator and Parent/Guardian based on maturity level of minor)

2.1.1.8 Willing to use acceptable forms of contraception, if applicable, or abstinence to prevent pregnancy.

EXCLUSION CRITERIA:

2.1.1.9 Any of the following hematologic abnormalities

* Hemoglobin less than 10.0 g/dL
* Neutrophil count less than 1500/mm(3)
* Platelet count less than 75,000/mm(3)
* Prothrombin time (PT) or partial thromboplastin time (PTT) greater than or equal to 1.5 times upper limits of normal (ULN) (with the exception of patients with known clotting disorders or known lupus anticoagulant).

2.1.1.10 Any of the following hepatic abnormalities

* Alanine transaminase (ALT)/ serum glutamate-pyruvate transaminase (SGPT) and/or Aspartate aminotransferase (AST)/Serum glutamic oxaloacetic transaminase (SGOT) greater than 2.5 times ULN
* Total bilirubin greater than 1.5 times ULN unless attributable to protease inhibitor therapy.

2.1.1.11 Positive tests (antibody and/or antigen) for hepatitis B and hepatitis C viruses, unless the result is consistent with prior vaccination or prior infection with full recovery.

2.1.1.12 Acute infection requiring therapy at time of enrollment. Participants may be eligible for study after being on stable and appropriate anti-infective therapy.

2.1.1.13 Chemotherapy for active cancer.

2.1.1.14 Documented history of non-adherence to antiretroviral treatment regimen within 12 months of study entry.

2.1.1.15 Pregnancy or breastfeeding.

2.1.1.16 Use of immunosuppressive or immunomodulating agents within 8 weeks of study enrollment. Note: patients receiving oral corticosteroids for management of asthma or contact hypersensitivity for less than or equal to 14 days in duration will be allowed to enroll as long as it has been greater than or equal to 30 days since oral corticosteroid administration.

2.1.1.17 Known immediate hypersensitivity to yeast or any of the vaccine components.

2.1.1.18 Use of investigational agents within 4 weeks prior to study enrollment.

2.1.1.19 Active external genital warts requiring treatment or cervical intraepithelial neoplasia (CIN)2/3

2.1.1.20 Any clinically significant diseases (other than HIV infection) or findings during study screening that, in the opinion of the Principal Investigator or Lead Associate Investigator, may interfere with the study.

Cohort 2 Inclusion and Exclusion Eligibility Criteria:

Inclusion Criteria

2.1.2.1 Age 12 to 26 years

2.1.2.2 Females and males

2.1.2.3 HIV-positive

2.1.2.4 CD4 cell count and HIV-1 RNA level parameters

* CD4 cell count greater than or equal to 500 cells/mm(3)
* HIV-1 RNA level by RT PCR less than or equal to 20,000 copies/ml.

2.1.2.5 Not receiving antiretroviral treatment with CD4 and viral load parameters as outlined in 2.1.2.4.

2.1.2.6 Patients greater than or equal to 18 years willing to provide informed consent or parent/guardian willing to provide informed consent for minor children less than 18 years of age.

2.1.2.7 Informed assent for patients 12-17 years of age (Optional at the discretion of the Principal Investigator and Parent/Guardian based on maturity level of minor)

2.1.2.8 Willing to use acceptable forms of contraception, if applicable, or abstinence to prevent pregnancy.

EXCLUSION CRITERIA:

2.1.2.9 Any of the following hematologic abnormalities:

* Hemoglobin less than 10.0 g/dL
* Neutrophil count less than 1500/mm(3)
* Platelet count less than 75,000/mm(3)
* PT or PTT greater than or equal to 1.5 times ULN (with the exception of patients with known clotting disorders or known lupus anticoagulant).

2.1.2.10 Any of the following hepatic abnormalities

* ALT/SGPT and/or AST/SGOT greater than 2.5 times ULN
* Total bilirubin greater than 1.5 times ULN unless attributable to protease inhibitor therapy.

2.1.2.11 Positive tests (antibody and/or antigen) for hepatitis B and hepatitis C viruses, unless the result is consistent with prior vaccination or prior infection with full recovery.

2.1.2.12 Acute infection requiring therapy at time of enrollment. Participants may be eligible for study after being on stable and appropriate anti-infective therapy.

2.1.2.13 Chemotherapy for active cancer.

2.1.2.14 Pregnancy or breastfeeding.

2.1.2.15 Use of immunosuppressive or immunomodulating agents within 8 weeks prior to study enrollment. Note: patients receiving oral corticosteroids for management of asthma or contact hypersensitivity for less than or equal to 14 days in duration will be allowed to enroll as long as it has been greater than or equal to 30 days since oral corticosteroid administration.

2.1.2.16 Known immediate hypersensitivity to yeast or any of the vaccine components.

2.1.2.17 Use of investigational agents within 4 weeks prior to study enrollment.

2.1.2.18 Active external genital warts requiring treatment or CIN2/3

2.1.2.19 Any clinically significant diseases (other than HIV infection) or findings during study screening that, in the opinion of the Principal Investigator or Lead Associate Investigator may interfere with the study.

Cohort 3 Inclusion and Exclusion Eligibility Criteria:

INCLUSION CRITERIA:

2.1.3.1 Age 12 to 26 years

2.1.3.2 Females and males

2.1.3.3 HIV-negative

2.1.3.4 Patients greater than or equal to 18 years willing to provide informed consent or parent/guardian willing to provide informed consent for minor children less than 18 years of age.

2.1.3.5 Informed assent for patients 12-17 years of age (Optional at the discretion of the Principal Investigator and Parent/Guardian based on maturity level of minor)

2.1.3.6 Willing to use acceptable forms of contraception, if applicable, or abstinence to prevent pregnancy.

EXCLUSION CRITERIA:

2.1.3.7 Any of the following hematologic abnormalities:

* Hemoglobin less than 10.0 g/dL
* Neutrophil count less than 1500/mm(3)
* Platelet count less than 75,000/mm(3)
* PT or PTT greater than or equal to 1.5 times ULN (with the exception of patients with known clotting disorders or known lupus anticoagulant).

2.1.3.8 Any of the following hepatic abnormalities

* ALT/SGPT and/or AST/SGOT greater than 2.5 times ULN
* Total Bilirubin greater than 1.5 times ULN unless attributable to protease inhibitor therapy.

2.1.3.9 Positive tests (antibody and/or antigen) for HIV, hepatitis B and hepatitis C viruses, unless the result is consistent with prior vaccination or prior infection with full recovery.

2.1.3.10 Acute infection requiring therapy at time of enrollment. Participants may be eligible for study after being on stable and appropriate anti-infective therapy.

2.1.3.11 Chemotherapy for active cancer.

2.1.3.12 Pregnancy or breastfeeding

2.1.3.13 Use of immunosuppressive or immunomodulating agents within 8 weeks prior to study enrollment. Note: patients receiving oral corticosteroids for management of asthma or contact hypersensitivity for less than or equal to 14 days in duration will be allowed to enroll as long as it has been greater than or equal to 30 days since oral corticosteroid administration.

2.1.3.14 Known immediate hypersensitivity to yeast or any of the vaccine components.

2.1.3.15 Use of investigational agents within 4 weeks prior to study enrollment.

2.1.3.16 Active external genital warts requiring treatment or carcinoma in-situ 2/3 (CIN2/3)

2.1.3.17 Any clinically significant diseases or findings during study screening that, in the opinion of the Principal Investigator or Lead Associate Investigator may interfere with the study.

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2009-06-29 (Actual); Primary Completion 2012-09-22 (Actual); Study Completion 2013-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoyoung M Maeng, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Background] Koutsky LA, Galloway DA, Holmes KK. Epidemiology of genital human papillomavirus infection. Epidemiol Rev. 1988;10:122-63. doi: 10.1093/oxfordjournals.epirev.a036020. PMID 2852116
- [Background] Munoz N, Bosch FX, de Sanjose S, Herrero R, Castellsague X, Shah KV, Snijders PJ, Meijer CJ; International Agency for Research on Cancer Multicenter Cervical Cancer Study Group. Epidemiologic classification of human papillomavirus types associated with cervical cancer. N Engl J Med. 2003 Feb 6;348(6):518-27. doi: 10.1056/NEJMoa021641. PMID 12571259
- [Background] Koshiol JE, Laurent SA, Pimenta JM. Rate and predictors of new genital warts claims and genital warts-related healthcare utilization among privately insured patients in the United States. Sex Transm Dis. 2004 Dec;31(12):748-52. doi: 10.1097/01.olq.0000145851.76025.ad. PMID 15608590
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0024.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in Cohort 2 - 0.5 mL dose injected intramuscular (IM) group.
Groups:
- Cohort 1 -.5 mL Dose Injected Intramuscular (IM): 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0
  Gardasil: 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months
  Survey: Administration of online risk behavior and knowledge survey done at week 0.
  Human immunodeficiency virus (HIV) positive, cluster of differentiation 4 (CD4) cell count > 350 cells/mm^3, Human immunodeficiency virus type 1 (HIV-1) Ribonucleic acid (RNA) level by reverse transcription-polymerase chain reaction (RT PCR) <20,000
- Cohort 3 -.5 mL Dose Injected Intramuscular (IM): 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0
  Gardasil: 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months
  Survey: Administration of online risk behavior and knowledge survey done at week 0.
  Healthy, Human immunodeficiency virus (HIV)-negative controls
Period: Overall Study
Arm/Group | Cohort 1 -.5 mL Dose Injected Intramuscular (IM) | Cohort 3 -.5 mL Dose Injected Intramuscular (IM)
Started | 8 | 18
Completed | 0 | 0
Not Completed | 8 | 18
Not completed — Lost to Follow-up | 1 | 10
Not completed — Study closing | 7 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Screen failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM): 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0
  Gardasil: 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months
  Survey: Administration of online risk behavior and knowledge survey done at week 0.
  Human immunodeficiency virus (HIV) positive, cluster of differentiation 4 (CD4) cell count > 350 cells/mm^3, Human immunodeficiency virus type 1 (HIV-1) Ribonucleic acid (RNA) level by reverse transcription-polymerase chain reaction (RT PCR) <20,000
- Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM): 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0
  Gardasil: 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months
  Survey: Administration of online risk behavior and knowledge survey done at week 0.
  Healthy, Human immunodeficiency virus (HIV)-negative controls
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM) | Total
Number analyzed (Participants) | 8 | 18 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 9
  Between 18 and 65 years | 4 | 13 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.68 (3.9) | 20.86 (5.1) | 20.19 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 12
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 16 | 23
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 5 | 12 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 18 | 26

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity of the Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine in Human Immunodeficiency Virus (HIV)-Infected Preadolescents, Adolescents and Young Adults 12-26 Years of Age
Description: Immunogenicity was measured by the vaccine-induced antibody response collectively for preadolescents, adolescents and young adults an reported per cohort for participants with HIV and without HIV. Participants' serum was used to check the level of human papillomavirus (HPV) neutralization antibody. Neutralizing antibody is an antibody that can bind to the infectious organism such as viruses and stop the spread of the disease. The antibody level was compared between the participants with HIV and without HIV.
Time Frame: Up to 36 months
Population: No participants were analyzed at 48 months because they were all of study before month 48 and the study ended.
Measure: Geometric Mean (Full Range); unit: EU/ml
Arm/Group | Cohort 1 -.5 mL Dose Injected Intramuscular (IM) | Cohort 3 -.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 8 | 17
EU/ml
  HPV-6 at Baseline | NA [7 to 7] — Geometric mean is below the detectable limit (<7). | 12.24 [7 to 29]
  HPV-6 at 7 Months: number analyzed (Participants) | 8 | 15
  HPV-6 at 7 Months | 955.77 [275.2 to 3452] | 598.90 [89 to 3180]
  HPV-6 at 12 Months: number analyzed (Participants) | 8 | 14
  HPV-6 at 12 Months | 311.15 [34.4 to 3218] | 286.07 [43 to 1670]
  HPV-6 at 24 Months: number analyzed (Participants) | 7 | 9
  HPV-6 at 24 Months | 280.22 [62.19 to 2058] | 186.13 [68 to 694]
  HPV-6 at 36 Months: number analyzed (Participants) | 5 | 3
  HPV-6 at 36 Months | 189.82 [63.14 to 1417] | 169.78 [57 to 504]
  HPV-6 at 48 Months: number analyzed (Participants) | 0 | 0
  HPV-11 at Baseline | 7.00 [7 to 7] | 14.61 [7 to 29]
  HPV-11 at 7 Months: number analyzed (Participants) | 8 | 15
  HPV-11 at 7 Months | 1873.68 [677.6 to 9992] | 1159.81 [165 to 3937]
  HPV-11 at 12 Months: number analyzed (Participants) | 8 | 14
  HPV-11 at 12 Months | 611.98 [85.85 to 5620] | 457.23 [145 to 2195]
  HPV-11 at 24 Months: number analyzed (Participants) | 7 | 9
  HPV-11 at 24 Months | 477.21 [137.4 to 2806] | 232.88 [91 to 732]
  HPV-11 at 36 Months: number analyzed (Participants) | 7 | 3
  HPV-11 at 36 Months | 285.92 [100.8 to 1997] | 171.53 [81 to 401]
  HPV-11 at 48 Months: number analyzed (Participants) | 0 | 0
  HPV-16 at Baseline | NA [7 to 7] — Geometric mean is below the detectable limit (<7). | 12.24 [7 to 29]
  HPV-16 at 7 Months: number analyzed (Participants) | 8 | 15
  HPV-16 at 7 Months | 1943 [424.6 to 9273] | 2876 [601.13 to 18831.61]
  HPV-16 at 12 Months: number analyzed (Participants) | 8 | 14
  HPV-16 at 12 Months | 523.7 [71.67 to 3745] | 1155 [286.08 to 14845.00]
  HPV-16 at 24 Months: number analyzed (Participants) | 7 | 9
  HPV-16 at 24 Months | 359.7 [43.05 to 1462] | 665 [148.01 to 6428.56]
  HPV-16 at 36 Months: number analyzed (Participants) | 5 | 3
  HPV-16 at 36 Months | 295 [47.19 to 1132] | 611 [211.49 to 5401.17]
  HPV-16 at 48 Months: number analyzed (Participants) | 0 | 0
  HPV-18 at Baseline | 7.00 [7 to 7] | 8.04 [7 to 168]
  HPV-18 at 7 Months: number analyzed (Participants) | 8 | 15
  HPV-18 at 7 Months | 1453.32 [424.6 to 9273] | 1171.10 [201 to 9659]
  HPV-18 at 12 Months: number analyzed (Participants) | 8 | 14
  HPV-18 at 12 Months | 409.57 [71.67 to 3745] | 478.98 [77 to 8920]
  HPV-18 at 24 Months: number analyzed (Participants) | 7 | 9
  HPV-18 at 24 Months | 253.70 [43.05 to 1462] | 301.76 [101 to 2856]
  HPV-18 at 36 Months: number analyzed (Participants) | 5 | 3
  HPV-18 at 36 Months | 202.29 [47.19 to 1132] | 289.66 [97 to 1756]
  HPV-18 at 48 Months: number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Human Papilloma Virus (HPV) Vaccine Immunogenicity Between Human Immunodeficiency Virus (HIV)-Infected Participants Receiving Highly Active Antiretroviral Therapy (HAART) & Those Not Receiving HAART With Similar T-lymphocytes (CD4) & Viral Load Parameters
Description: Match per the HIV level at study entry to compare between cohort 1 and 2.
Time Frame: At study entry
Population: This outcome measure was not done because no participants were enrolled in Cohort 2 - 0.5 mL dose injected intramuscular (IM) group.
Groups:
- Cohort 2 - 0.5 mL Dose Injected Intramuscular (IM): 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0.
  This outcome measure was to be done in cohort 2 only but no participants were enrolled in Cohort 2 - 0.5 mL dose injected intramuscular (IM) group.
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 2 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Log Change in Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Levels After Human Papilloma Virus (HPV) Vaccination
Description: Within each cohort, the number of participants with a change in log^10 HIV-1 RNA levels will be determined between day 1 and day 7 and will be evaluated to see if the values at the two time points are not statistically different from one another. HIV-1 RNA levels below the lower limits of detection (50 copies/ml) will be expressed as 1.69 log^10 on a logarithmic scale equivalent to 49 copies/ml. There is at least 95% power to detect a change from day 1 to day 7 with an effect size of 1 standard deviation (SD) and a 0.025 two-sided alpha level test (0.05/2 cohorts) after allowing for a Bonferroni adjustment.
Time Frame: Baseline, and months 1, 3, 7 and 12
Population: Only Cohort 1 is applicable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 8
Participants
  Baseline | 1
  1 Month | NA — HIV RNA was undetectable or lower than baseline.
  3 Months | NA — HIV RNA was undetectable or lower than baseline.
  7 Months | 1
  12 Months | NA — HIV RNA was undetectable or lower than baseline.

4. Secondary Outcome: Fold Change in Anti-Human Papilloma Virus (HPV) Titer and T-lymphocytes (CD4) Count (Only at Baseline)
Description: Fold change in anti-HPV titer with baseline T-lymphocytes (CD4) count. Fold change is a measure of the antibody titer after vaccination divided by the baseline titer.
Time Frame: Months 7, 12, 24 and 36
Population: A different number of samples were available for the assay at 7, 12, 24 and 36 months as noted in the table.
Measure: Median (Full Range); unit: Fold Change
Units Other Than Participants: Blood Samples
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 8 | 14
Number analyzed (Blood Samples) | 8 | 14
Fold Change
  anti-HPV-6 at 7 months | 142.64 [39.32 to 493.10] | 90.22 [12.65 to 432.46]
  anti-HPV-6 at 12 months: number analyzed (Participants) | 8 | 13
  anti-HPV-6 at 12 months: number analyzed (Blood Samples) | 8 | 13
  anti-HPV-6 at 12 months | 42.00 [4.91 to 459.65] | 28.48 [6.08 to 223.17]
  anti-HPV-6 at 24 months: number analyzed (Participants) | 7 | 8
  anti-HPV-6 at 24 months: number analyzed (Blood Samples) | 7 | 8
  anti-HPV-6 at 24 months | 55.00 [8.88 to 293.98] | 18.35 [9.05 to 92.65]
  anti-HPV-6 at 36 months: number analyzed (Participants) | 5 | 3
  anti-HPV-6 at 36 months: number analyzed (Blood Samples) | 5 | 3
  anti-HPV-6 at 36 months | 16.70 [9.02 to 202.47] | 24.37 [8.13 to 67.37]
  anti-HPV-11 at 7 months | 235.69 [96.79 to 1427.45] | 189.84 [23.57 to 532.02]
  anti-HPV-11 at 12 months: number analyzed (Participants) | 8 | 13
  anti-HPV-11 at 12 months: number analyzed (Blood Samples) | 8 | 13
  anti-HPV-11 at 12 months | 68.90 [12.26 to 802.92] | 71.57 [6.58 to 296.64]
  anti-HPV-11 at 24 months: number analyzed (Participants) | 7 | 8
  anti-HPV-11 at 24 months: number analyzed (Blood Samples) | 7 | 8
  anti-HPV-11 at 24 months | 69.29 [19.63 to 400.79] | 37.47 [4.92 to 98.87]
  anti-HPV-11 at 36 months: number analyzed (Participants) | 5 | 3
  anti-HPV-11 at 36 months: number analyzed (Blood Samples) | 5 | 3
  anti-HPV-11 at 36 months | 23.69 [14.40 to 285.29] | 22.22 [11.57 to 54.14]
  anti-HPV-16 at 7 months | 589.91 [211.16 to 2978.10] | 382.60 [24.10 to 2690.23]
  anti-HPV-16 at 12 months | 183.15 [59.14 to 805.85] | 142.79 [9.84 to 2120.71]
  anti-HPV-16 at 24 months | 137.73 [40.47 to 437.20] | 59.87 [7.52 to 918.37]
  anti-HPV-16 at 36 months: number analyzed (Participants) | 6 | 3
  anti-HPV-16 at 36 months: number analyzed (Blood Samples) | 6 | 3
  anti-HPV-16 at 36 months | 78.30 [0.00 to 321.86] | 30.81 [20.34 to 250.89]
  anti-HPV-18 at 7 months | 145.36 [60.66 to 1324.73] | 142.60 [7.66 to 1379.84]
  anti-HPV-18 at 12 months: number analyzed (Participants) | 8 | 13
  anti-HPV-18 at 12 months: number analyzed (Blood Samples) | 8 | 13
  anti-HPV-18 at 12 months | 55.35 [10.24 to 535.03] | 39.58 [4.64 to 1274.25]
  anti-HPV-18 at 24 months: number analyzed (Participants) | 7 | 8
  anti-HPV-18 at 24 months: number analyzed (Blood Samples) | 7 | 8
  anti-HPV-18 at 24 months | 36.63 [6.15 to 208.86] | 22.46 [3.28 to 408.05]
  anti-HPV-18 at 36 months: number analyzed (Participants) | 5 | 3
  anti-HPV-18 at 36 months: number analyzed (Blood Samples) | 5 | 3
  anti-HPV-18 at 36 months | 94.24 [10.00 to 161.72] | 20.34 [13.88 to 250.89]

5. Secondary Outcome: T-lymphocytes (CD4) Count (Only at Baseline)
Description: Baseline T-lymphocytes (CD4) count.
Time Frame: Baseline
Measure: Median (Full Range); unit: Cells/mm^3
Units Other Than Participants: Blood Samples
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 8 | 14
Number analyzed (Blood Samples) | 8 | 14
Cells/mm^3 | 643 [457 to 1232] | 753 [425 to 2041]

6. Secondary Outcome: Number of Participants With Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) Positivity by Oral/Buccal Swabs at Baseline in the Study Cohort Populations
Description: Human papillomavirus (HPV) deoxyribonucleic acid (DNA) positivity by oral/buccal swabs was performed by swabbing the oral/buccal mucosa and
Time Frame: Baseline
Population: Data not collected.
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Human Papillomavirus (HPV) Deoxyribonucleic Acid (DNA) Positivity by Anogenital Swabs
Description: HPV DNA positivity by anogenital swabs was performed by Papanicolaou test (PAP) test. PAPs were not conducted when the participant stated that she was not sexually active.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 8 | 18
Participants | 2 | 10

8. Secondary Outcome: Number of Participants Who Completed The Youth Risk Behavior Surveillance System (YRBSS)
Description: Here are the number of participants who properly completed (i.e., answered correctly) the YRBSS. The human papilloma virus (HPV) & human immunodeficiency virus (HIV) knowledge and risk and sexual behaviors was assessed by a middle school or high school version of web-based Youth Risk Behavior Survey developed by Centers for Disease Control and Prevention (CDC). The Youth Risk Behavior Surveillance System (YRBSS) developed by the CDC was used to monitor six categories of priority health risk behaviors among middle school and high school youth: behaviors that contribute to unintentional injuries and violence; tobacco use; alcohol and other drug use; sexual behaviors that contribute to unintended pregnancy and sexually transmitted diseases (STDs), including human immunodeficiency virus (HIV) infections; unhealthy dietary behaviors; and physical inactivity and determine the number of participants who answered correctly on the assessment tool (i.e., YRBSS).
Time Frame: Baseline
Population: Participant data is combined for this outcome measure as pre-specified by the protocol. No statistical comparisons between cohorts were planned.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants in Cohort 1 and Cohort 3. Cohort 1 - 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0 Gardasil: 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months Survey: Administration of online risk behavior and knowledge survey done at week 0.
  Human immunodeficiency virus (HIV) positive, cluster of differentiation 4 (CD4) cell count > 350 cells/mm^3, Human immunodeficiency virus type 1 (HIV-1) Ribonucleic acid (RNA) level by reverse transcription-polymerase chain reaction (RT PCR) <20,000.
  Cohort 3 - 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months (+/- 2 weeks) and knowledge survey at week 0 Gardasil: 0.5 mL dose injected intramuscular (IM) at 0, 2 and 6 months Survey: Administration of online risk behavior and knowledge survey done at week 0.
  Healthy, Human immunodeficiency virus (HIV)-negative controls
Arm/Group | All Participants
Number analyzed (Participants) | 26
Participants | 26

9. Secondary Outcome: Number of Participants With Serum for Human Papilloma Virus (HPV) Antibody Titers Performed by Merck (Competitive Luminex Assay)
Description: Participants collection Tube: 10ml red top tube (RTT) send via courier to National Cancer Institute (NCI) FCRF for processing, aliquoting and cryopreservation by Baselar lab. Batched specimens to be sent to Merck for HPV antibody titers.
Time Frame: 0, 1, 2, 3, 6, 7, 12, 18, 24, 30, 36, 42, and 48 hours
Population: The lab assigned to do this assay was not able to perform the study.
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Functional Human Papilloma Virus (HPV) Antibody Neutralization Assays
Description: Month 7 anti-HPV Ab titer was correlated with Neutralization Assay (PBNA) antibody titers and analyzed by the secreted alkaline phosphatase (SEAP)/enzyme-linked immunosorbent assay (ELISA) R.
Time Frame: At 7 months
Population: 15/18 participants were analyzed in Cohort 3 because one participant was a screen failure, one participant withdrew from study and one participant was taken off study.
Measure: Number; unit: Coefficient
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 8 | 15
Coefficient
  HPV-16 | 0.90476 | 0.81071
  HPV-18 | 0.97619 | 0.88571
Statistical Analysis 1: Comparison: Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM); Test type: Other; p = 0.0020, Spearman correlation (non-parametric) — The reported p-value is representative of the changes in HPV-16 at 7 months in Cohort 1
Statistical Analysis 2: Comparison: Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM); Test type: Other; p < .0001, Spearman correlation (non-parametric) — The reported p-value is representative of the changes in HPV-18 at 7 months in Cohort 1
Statistical Analysis 3: Comparison: Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM); Test type: Other; p = 0.0002, Spearman correlation (non-parametric) — The reported p-value is representative of the changes in HPV-16 at 7 months in Cohort 2
Statistical Analysis 4: Comparison: Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM); Test type: Other; p < .0001, Spearman correlation (non-parametric) — The reported p-value is representative of the changes in HPV-18 at 7 months in Cohort 2

11. Secondary Outcome: Cryopreserved Peripheral Blood Mononuclear Cells (PBMCs) for Human Papilloma Virus (HPV) & Human Immunodeficiency Virus (HIV) Lymphocyte Proliferation Assays, Cytokine Induction Assay, Luminex Multi-cytokine Profiling of PBMCs
Description: Participants collection tube: 6 tubes sodium heparin 10ml green top tube (GTT) (60ml total) send via courier to National Cancer Institute (NCI) FCRF for processing, aliquoting and cryopreservation by Baselar lab according to protocol provided by the investigator. Note: HIV lymphocyte proliferation assays will only be performed in HIV-infected subjects
Time Frame: 0, 1, 3, 7, 12, 24, 36, and 48 hours
Population: Samples were not available to perform the study. This type of immune assay requires a large number of PBMCs in pairs including baseline samples, but the collection was inadequate for the assay and the assay was not done.
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Extended Fluorescence Activated Cell Sorting (FACS)/Quantitative Lymphocyte Subpopulation Studies
Description: Extended FACS/Quantitative lymphocyte subpopulation studies human immunodeficiency virus (HIV)-infected subjects only (Cohorts 1 and 2) using a 10ml sodium heparin green top tube (GTT).
Time Frame: 0, 1, 3, 7, 12, 18, 24, 30, 36, 42, and 48 hours
Population: Samples were not available to perform the study. This type of immune assays requires a large number of PBMCs in pairs including baseline samples, but the collection was inadequate for the assay and the assay was not done.
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Quantitative Measurement of Human Immunodeficiency Virus (HIV)-Related Chemokines Macrophage Inflammatory Proteins (MIP)-1 Alpha (α), MIP-1 Beta (β) and Regulated Upon Activation, Normal T Cell Expressed and Presumably Secreted (RANTES)
Description: Collection tube: 10ml red top tube (RTT) send via courier to National Cancer Institute (NCI) FCRF for processing, aliquoting and cryopreservation by Baselar lab.
Time Frame: 0, 1, 2, 3, 6, 7, 12, 18, 24, 30, 36, 42, and 48 hours
Population: This outcome measure was not done because there were not enough samples available to do a series (e.g., multiple timepoints).
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Cryopreserved Whole Blood for Human Papilloma Virus (HPV) Deoxyribonucleic Acid (DNA) Testing
Description: Three collection tube: 6ml purple top ethylenediamine tetraacetic acid (EDTA) tubes (18ml total)
Time Frame: 0, 7, 12, 24, 36, and 48 Months
Population: Data not collected.
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Research Assays Immunologic Responses for Human Immunodeficiency Virus (HIV) Infected Subjects Only
Description: Two collection tubes: 10ml sodium heparin green top tube (GTT) (20ml total) from HIV infected subjects only (Cohorts 1 and 2).
Time Frame: Month 0 only
Population: Data not collected.
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, up to 43 months and 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
Number analyzed (Participants) | 8 | 18
Participants | 8 | 16

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, up to 43 months and 8 days.
Arm/Group | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/18
Other Adverse Events (participants affected / at risk) | 8/8 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) (N=8) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM) (N=18)
Infection with unknown absolute neutrophil count (ANC): Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Pain: Abdomen Not Otherwise Specified (NOS) (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 0.5 mL Dose Injected Intramuscular (IM) (N=8) | Cohort 3 - 0.5 mL Dose Injected Intramuscular (IM) (N=18)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 7 (11) | 3 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (7) | 4 (4)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (2) | 2 (7)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 4 (7) | 4 (7)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dermatology/Skin - Other (Lesion) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatology/Skin - Other (Macular eruption) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatology/Skin - Other (Papulopustular eruption) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Wart) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 3 (4)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 0 (0)
Flu-like syndrome (General disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 1 (3) | 0 (0)
Hemorrhage, GU::Vagina (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection - Other (Flu) (Infections and infestations) | 1 (1) | 1 (1)
Infection - Other (H1N1 influenza) (Infections and infestations) | 1 (1) | 0 (0)
Infection - Other (Herpes) (Infections and infestations) | 0 (0) | 1 (3)
Infection - Other (Upper airway NOS) (Infections and infestations) | 0 (0) | 1 (2)
Infection - Other (Upper airway strep infection) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lip/perioral (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Middle ear (otitis media) (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pharynx (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Soft tissue NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Vagina (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Middle ear (otitis media) (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Skin (cellulites) (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 1 (1) | 1 (1)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (3)
Infection with unknown ANC::Vagina (Infections and infestations) | 0 (0) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 5 (13) | 10 (22)
Insomnia (General disorders) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (4) | 4 (6)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 4 (6)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 3 (5) | 5 (6)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (6) | 1 (3)
Ocular/Visual - Other (Linear visual field deficit OS) (Eye disorders) | 1 (1) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 2 (3) | 3 (3)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (7)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Supraventricular and nodal arrhythmia::Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight loss (General disorders) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT00798265/Prot_SAP_000.pdf
  • Informed Consent Form (2011-06-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT00798265/ICF_001.pdf